CLINICAL TRIAL: NCT05238597
Title: A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled Clinical Trial Evaluating the Safety, Tolerability, and Efficacy of A197 in Subjects With Dry Eye Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of A197 in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aramis Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A197-CS-201
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A197 Ophthalmic Solution, High Dose (Experimental)
  Interventions: Drug: A197 Ophthalmic Solution
- A197 Ophthalmic Solution, Low Dose (Experimental)
  Interventions: Drug: A197 Ophthalmic Solution
- A197 Vehicle Control (Placebo Comparator)
  Interventions: Drug: A197 Vehicle Control
- Active Comparator (Active Comparator)
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: A197 Ophthalmic Solution — A197 Ophthalmic Solution
  Arms: A197 Ophthalmic Solution, High Dose; A197 Ophthalmic Solution, Low Dose
Drug: A197 Vehicle Control — A197 Vehicle Control
  Arms: A197 Vehicle Control
Drug: Active Comparator — Active Comparator
  Arms: Active Comparator

SUMMARY:
The objectives of this trial are to assess the safety, tolerability and efficacy of A197 ophthalmic solution in comparison to a vehicle control in the treatment of subjects with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any study-related assessments
* Have a history of Dry Eye Disease in both eyes for at least 12 months prior to Visit 1
* Willing and able to follow instructions and can be present for required study visits

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Use of topical ophthalmic medications, artificial tears, eye drops and gels in either eye
* Use of contact lenses within 90 days prior to Visit 1 and throughout the study
* Have had an ocular infection in either eye within 90 days prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total corneal fluorescein staining (CFS) | 12 Weeks
  Corneal Fluorescein Staining (tCFS) is graded based on a modified National Eye Institute (NEI) scale. The NEI scale divides the cornea in 5 regions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-4 using 0.5 unit increments; 0 corresponds to no staining, 4 corresponds to maximum staining. The total score is the sum of the 5 regions ranging from 0-20.

SECONDARY OUTCOMES:
Change from baseline in eye dryness via the Visual Analogue Scale (VAS) | 12 Weeks
  Eye dryness is rated on a visual analogue scale (VAS) ranging from 0-100; 0 corresponds to no symptoms and 100 to severe symptoms.
Change from baseline in lissamine green conjunctival staining (LGCS) | 12 Weeks
  Lissamine green conjunctival staining (LGCS) is graded based on the NEI Scale. The NEI scale divides the conjunctiva in 6 regions with the score for each region ranging from 0-3; 0 corresponds to no staining, 3 corresponds to maximum staining. The total score is the sum of the 6 regions ranging from 0-18.
Change from baseline in bulbar conjunctival hyperemia (CCLRU) | 12 Weeks
  Bulbar conjunctival hyperemia is graded based on the Cornea and Contact Lens Research Unit (CCLRU) grading scale where 0 corresponds to none, 4 corresponds to severe.

CONTACTS AND LOCATIONS:
Overall Officials: David S Tierney, MD, Study Director — Aramis Biosciences
Locations (24):
- United States (24):
  - Aramis Site 113, Birmingham, Alabama
  - Aramis Site 121, Garden Grove, California
  - Aramis Site 120, Glendale, California
  - Aramis Site 106, Long Beach, California
  - Aramis Site 124, Los Angeles, California
  - Aramis Site 107, Murrieta, California
  - Aramis Site 102, Newport Beach, California
  - Aramis Site 116, Petaluma, California
  - Aramis Site 109, Rancho Cordova, California
  - Aramis Site 101, Delray Beach, Florida
  - Aramis Site 112, Jacksonville, Florida
  - Aramis Site 117, Largo, Florida
  - Aramis Site 118, Edgewood, Kentucky
  - Aramis Site 114, Kansas City, Missouri
  - Aramis Site 111, St Louis, Missouri
  - Aramis Site 108, Las Vegas, Nevada
  - Aramis Site 110, Garner, North Carolina
  - Aramis Site 122, Shelby, North Carolina
  - Aramis Site 119, Mason, Ohio
  - Aramis Site 123, Cranberry Township, Pennsylvania
  - Aramis Site 115, Goodlettsville, Tennessee
  - Aramis Site 103, Memphis, Tennessee
  - Aramis Site 104, Lakeway, Texas
  - Aramis Site 105, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473